CLINICAL TRIAL: NCT06838208
Title: Efficacy and Safety of Tislelizumab Combined With Chemotherapy and Relayed Radiotherapy in the First-line Treatment of Extensive Small Cell Lung Cancer: a Prospective, Multicenter, Phase II Clinical Study
Brief Title: Tislelizumab Combined With Chemotherapy and Relayed Radiotherapy in First-line Treatment of ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shuanghu Yuan, Professor, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRAD1; CRTOG2501 (Other: CRTOG)
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-02

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tislelizumab; Carboplatin; Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab plus chemo and radiotherapy (Experimental): Experimental treatment
  1. Drug: Tislelizumab, Carboplatin /Cisplatin, Etoposide
     • Tislelizumab (200 mg IV Q3W) in combination with chemotherapy consisting of etoposide (100 mg/m² IV Days 1-3 of each 21-day cycle) and platinum (cisplatin 75 mg/m² IV Q3W or carboplatin area under the plasma or serum concentration-time curve (AUC) 5 IV Q3W) for 4 cycles. Then maintenance consists of Tislelizumab Q3W and will continue until disease progression, loss of clinical benefit, unacceptable toxicity, or withdrawal of informed consent，up to 2 years.
  2. Radiotherapy:
     * Induction therapy stage LDRT: lung lesions, 15Gy/5f;
     * Maintenance therapy phase SBRT: The main residual lesions evaluated by the investigators, 30Gy/5f；
  Control group: This study refers to the Phase III RATIONALE-312 study, the reported median PFS was 4.7 months in patients treated with Tislelizumab combined with chemotherapy. This regimen has been recommened as 1L treatment for ES-SCLC in the CSCO guidelines.
  Interventions: Drug: Tislelizumab, Carboplatin /Cisplatin, Etoposide

INTERVENTIONS:
Drug: Tislelizumab, Carboplatin /Cisplatin, Etoposide — Induction therapy stage LDRT: lung lesions, 15Gy/5f; Maintenance therapy phase SBRT: The main residual lesions evaluated by the investigators, 30Gy/5f；
  Other Names: radiotherapy

SUMMARY:
To explore the efficacy and safety of Tislelizumab combined with chemotherapy and relayed radiotherapy in the first-line treatment of extensive small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old, male or female, signed Informed Consent Form (ICF);
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
3. Histologically or cytologically confirmed ES-SCLC;
4. No prior systemic treatment for ES-SCLC;
5. At least one measurable (RECIST 1.1) chest lesion capable of 15Gy/5f irradiation;
6. Adequate hematologic and end organ function;

Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled, untreated brain metastasis;
2. Prior therapy with an antibody or drug against immune checkpoint pathways, including but not limited to, anti program death receptor-1 (anti-PD-1), anti-PD-L1, or anti cytotoxic T lymphocyte associated antigen 4 (anti CTLA-4) antibody;
3. Was administered a live vaccine ≤ 4 weeks before treatment;
4. Active autoimmune diseases or history of autoimmune diseases that may relapse;
5. Any condition that required systemic treatment with either corticosteroids or other immunosuppressive medication ≤ 14 days before treatment;
6. With a history of interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases;
7. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy within 2 weeks prior to treatment, including but not limited to tuberculosis infection;
8. Received therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to starting treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Baseline until PD or death, whichever occurs first or up to approximately 23 months
  To evaluate the efficacy of Tislelizumab + cisplatin or carboplatin + etoposide and radiotherapy in the intent to treat (ITT) Analysis Set as measured by investigator assessed progression free survival (PFS) according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until partial response (PR) or complete response (CR), whichever occurs or up to approximately 23 months
  To evaluate the efficacy of Tislelizumab + cisplatin or carboplatin + etoposide +radiotherapy in the ITT Analysis Set as measured by investigator assessed overall response rate (ORR), according to RECIST v1.1
Duration Of Response (DOR) | Baseline until partial response (PR) or complete response (CR), whichever occurs first, or up to approximately 23 months
  To evaluate the efficacy of Tislelizumab + cisplatin or carboplatin + etoposide+ radiotherapy in the ITT Analysis Set as measured by investigator assessed duration of response (DOR) according to RECIST v1.1
Disease Control Rate (DCR) | up to approximately 23 months
  To evaluate the efficacy of Tislelizumab + cisplatin or carboplatin + etoposide + radiotherapy in the ITT Analysis Set as measured by investigator assessed disease control rate (DCR) according to RECIST v1.1
6-moth/1-year Progression Free Survival (PFS) Rate | up to approximately 23 months
  The PFS rate will be defined as the proportion of participants free from PFS events at 6 month and 1st year after the first dose.
1-year Overall Survival (OS) rate | up to approximately 23 months
  The OS rate will be defined as the proportion of participants free from OS events at 1st year after the first dose.
Number Of Participants Experiencing Treatment-Emergent Adverse Events | up to approximately 23 months
  Incidence and severity of treatment-emergent adverse events (TEAEs) graded according to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Cancer Hospital, Hefei, Anhui, China